CLINICAL TRIAL: NCT01218048
Title: Phase II Study of Neoadjuvant Immune Biomarker Modulation With Cetuximab Followed by Adjuvant Therapy With Concurrent Chemoradiotherapy or Radiotherapy With or Without Cetuximab for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: ERBITUX® Followed by Adjuvant Treatment With Chemoradiation and ERBITUX® for Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Ferris (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Robert Ferris, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 08-013
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Carcinoma; Head and Neck; Cetuximab; Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma | interventions — Cetuximab; Surgical Procedures, Operative; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neo-Adjuvant Cetuximab (Experimental): Neo-Adjuvant Cetuximab + Surgery + Post-Surgical Radiation + Cisplatin (or Carboplatin)
  NOTE: Based the results of surgery if the treating physician feels patient is not a candidate for chemotherapy, radiation can be given alone or with cetuximab.
  Interventions: Drug: Cetuximab; Procedure: Surgery; Radiation: Post-surgical radiation; Drug: Cisplatin or carboplatin

INTERVENTIONS:
Drug: Cetuximab — Pre-Surgery: IV, 400 mg/m2 day 1 then 250 mg/m2 alone days 8 and 15; Post-surgery: IV, 250 mg/m2 weekly concurrent with RT
  Other Names: ERBITUX®
Procedure: Surgery — Surgery for tumor
Radiation: Post-surgical radiation — Radiation (2 Gy/d) to min of 60 Gy + max of 66 Gy post-surgery
Drug: Cisplatin or carboplatin — Cisplatin 30 mg/m2 or carboplatin AUC 1.5-2/week weekly, Concurrent with radiotherapy

SUMMARY:
There are currently no useful tests to identify patients who will respond to cetuximab therapy, notably because EGFR levels do not correlate with the clinical responses observed. Thus, the investigators are investigating the role of cellular immunity and immune escape mechanisms to explain the differential clinical response to cetuximab.

DETAILED DESCRIPTION:
This prospective phase II clinical trial of preoperative, single-agent cetuximab treated patients is being conducted in order to obtain specimens before and after 4 weeks of cetuximab for immune biomarker studies. Stage III/IV HNC patients will be treated with definitive surgical resection and observed for disease recurrence. Cetuximab will be administered for a 3-4 week preoperative period to study biomarker modulation in correlation clinical response by CT scan and tumor apoptosis/proliferation after tumor excision, immediately after neoadjuvant cetuximab but before surgery. We will biopsy the skin/acneiform rash in all patients to correlate rash with biomarker modulation and clinical response. Cetuximab may also be given in the adjuvant setting. A primary scientific hypothesis will be tested: does short term pre-operative exposure to cetuximab modulate blood immune biomarkers and is immune modulation associated with anti-tumor effect? Forty (n=40) patients with complete specimens (tumor, peripheral blood mononuclear cells (PBMC) and serum) are necessary to enable adequate statistical power to be reached using paired specimens. A secondary set of hypotheses will evaluate the association between pre-operative biomarker levels and modulation with disease recurrence. The proposed trial will accrue stage II, III or IV surgical candidates without distant metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, previously untreated HNC. Clinical stage III or IVA disease without distant metastases as determined by CT, and as defined by the American Joint Committee on Cancer Staging System, Sixth edition (See Appendix I).
* Primary tumors of the oral cavity, oropharynx, hypopharynx, or larynx will be included. Primary tumors of the sinuses, paranasal sinuses, or nasopharynx, or unknown primary tumors are NOT allowed.
* Macroscopic complete resection of the primary tumor must be planned.
* Age greater than or equal to 18 years.
* ECOG performance status 0-1.
* Adequate hematologic, renal and hepatic function, as defined by:

  * Absolute neutrophil count (ANC) greater than or equal to 1,500/ul, platelets greater than or equal to 100,000/ul.
  * Creatinine clearance > 40
  * Bilirubin less than or equal to 1.5 x ULN, AST or ALT less than or equal to 2.5 x ULN.
* Have signed written informed consent.

Exclusion Criteria:

* Subjects who fail to meet the above criteria.
* Prior severe infusion reaction to a monoclonal antibody.
* Pregnancy or breastfeeding. Women of childbearing potential (WOCBP) must practice acceptable methods of birth control to prevent pregnancy. Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.
* All WOCBP MUST have a negative pregnancy test within 7 days prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study. In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation. The Investigator must immediately notify BMS in the event of a confirmed pregnancy in a patient participating in the study.
* Subjects with an ECOG performance status of 2 or worse.
* Evidence of distant metastasis.
* Any other malignancy active within 5 years except for non-melanoma skin cancer or carcinoma in situ of the cervix, DCIS or LCIS of the breast.
* Prior history of HNC.
* Prior therapy targeting the EGFR pathway.
* Any unresolved chronic toxicity greater than or equal to grade 2 from previous anticancer therapy (except alopecia), according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
* Acute hepatitis, known HIV, or active uncontrolled infection.
* History of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, myocardial infarction within prior 6 months, untreated known coronary artery disease, uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Uncontrolled peptic or gastric ulcer disease, or gastrointestinal bleeding within prior 6 months.
* Active alcohol abuse or other illness that carries a likelihood of inability to comply with study treatment and follow-up.
* Treatment with a non-approved or investigational drug within 30 days prior to Day 1 of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2015-11-04 (Actual); Study Completion 2017-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rober L Ferris, MD, PhD, Principal Investigator — University of Pittsburgh Med Ctr (UPCI)
Locations (1):
- UPCI - Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Li J, Srivastava RM, Ettyreddy A, Ferris RL. Cetuximab ameliorates suppressive phenotypes of myeloid antigen presenting cells in head and neck cancer patients. J Immunother Cancer. 2015 Nov 17;3:54. doi: 10.1186/s40425-015-0097-6. eCollection 2015. PMID 26579227

RESULTS

PARTICIPANT FLOW:
Groups:
- Neo-Adjuvant Cetuximab: Patients with Head and Neck Squamous Cell Cancer (HNSCC) treated with Neo-Adjuvant Cetuximab + Surgery + Post-Surgical Radiation + Cisplatin (or Carboplatin)
  NOTE: Based the results of surgery if the treating physician feels patient is not a candidate for chemotherapy, radiation can be given alone or with cetuximab.
  Cetuximab: Pre-Surgery: IV, 400 mg/m^2 day 1 then 250 mg/m^2 alone days 8 and 15; Post-surgery: IV, 250 mg/m2 weekly concurrent with RT
  Post-surgical radiation: Radiation (2 Gy/d) to min of 60 Gy + max of 66 Gy post-surgery
  Cisplatin or carboplatin: Cisplatin 30 mg/m2 or carboplatin AUC 1.5-2/week weekly, Concurrent with radiotherapy
Period: Overall Study
Arm/Group | Neo-Adjuvant Cetuximab
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 58.6 [38 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: NK Cell Activation
Description: Cetuximab-mediated NK cell activation (percentage of activity) measures at pre-/post-cetuximab exposure for patients in peripheral blood lymphocytes (PBL) and tumor infiltrating lymphocytes (TIL) and in those patients that did and did not respond to treatment.
Time Frame: Prior to each weekly cetuximab treatment (up to 4 weeks); at the time of surgery (at 3-4 weeks after first cetuximab treatments)
Population: Participants that received preoperative treatment with single-agent cetuximab for a minimum of 3-4 weeks.Patients defined as responders, demonstrated upregulation of CD137 on tumor infiltrating NK cells following cetuximab therapy compared with non-responders.
Measure: Median (Inter-Quartile Range); unit: percentage of activity
Groups:
- Neo-Adjuvant Cetuximab: Patients with Head and Neck Squamous Cell Cancer (HNSCC) treated with Neo-Adjuvant Cetuximab + Surgery + Post-Surgical Radiation +/- Cisplatin (or Carboplatin): Intravenous Cetuximab (pre-surgery) 400 mg/m^2 alone days 8 and 15; then 250mg/m^2/week) for 3-4 weeks preoperatively, followed post-surgery by adjuvant chemoradiation with or without 250 mg/m^2 weekly cetuximab.
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 17
percentage of activity
  Percent NK cells (PBL): pre-cetuximab | 19 [13 to 22]
  Percent NK cells (PBL): post-cetuximab | 20 [12 to 27]
  Percent NK cells (TIL): pre-cetuximab | 4 [2 to 7]
  Percent NK cells (TIL): post-cetuximab | 3 [1 to 4]
  Percent CD16+ NK cells(PBL): pre-cetuximab | 55 [40 to 66]
  Percent CD16+ NK cells (PBL): post-cetuximab | 49 [34 to 65]
  Percent CD16+ NK cells (TIL): pre-cetuximab | 10 [4 to 15]
  Percent CD16+ NK cells (TIL): post-cetuximab | 6 [4 to 9]
  Percent Granzyme B+ cells (PBL): pre-cetuximab | 54 [46 to 66]
  Percent Granzyme B+ cells(PBL): post-cetuximab | 64 [54 to 71]
  Percent Granzyme B+ cells (TIL): pre-cetuximab | 17 [1 to 20]
  Percent Granzyme B+ cells (TIL): post-cetuximab | 21 [10 to 31]
  Percent Perforin+ cells (PBL): pre-cetuximab | 50 [42 to 68]
  Percent Perforin+ cells (PBL): post-cetuximab | 60 [46 to 78]
  Percent Perforin+ cells (TIL): pre-cetuximab | 6 [1 to 14]
  Percent Perforin+ cells (TIL): post-cetuximab | 10 [2 to 14]
  Percent CD107a+ cells (PBL): pre-cetuximab | 1 [0 to 4]
  Percent CD107a+ cells (PBL): post-cetuximab | 0 [0 to 0]
  Percent CD107a+ cells (TIL): pre-cetuximab | 36 [23 to 56]
  Percent CD107a+ cells (TIL): post-cetuximab | 60 [38 to 69]
  Percent CD137+ cells (PBL): pre-cetuximab | 2 [1 to 3]
  Percent CD137+ cells (PBL): post-cetuximab | 0 [0 to 0]
  Percent CD137+ cells (TIL): pre-cetuximab | 6 [3 to 10]
  Percent CD137+ cells (TIL): post-cetuximab | 10 [8 to 13]

2. Primary Outcome: Serum Cytokines Levels
Description: Serum cytokines levels measured at pre-/post-cetuximab, exposure measured in picogram per milliliter of plasma (pg/ml)
Time Frame: as for outcome 1
Population: Participants that received preoperative treatment with single-agent cetuximab for a minimum of 3-4 weeks.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 33
pg/ml
  Responders: pre-cetuximab GM-CSF | 2.5 [2.0 to 8.0]
  Non-responders: pre-cetuximab GM-CSF | 18.0 [2.0 to 22.0]
  Responders: post-cetuximab GM-CSF | 11.0 [7.0 to 13.0]
  Non-responders: post-cetuximab GM-CSF | 5.0 [2.0 to 12.5]
  Responders: pre-cetuximab CCL2 | 260 [175 to 500]
  Non-responders: pre-cetuximab CCL2 | 500 [100 to 1600]
  Responders: post-cetuximab CCL2 | 250 [200 to 400]
  Non-responders: post-cetuximab CCL2 | 200 [100 to 750]
  Responders: pre-cetuximab MP-1 alpha | 6.0 [5.0 to 9.5]
  Non-responders: pre-cetuximab MP-1 alpha | 10.0 [1.0 to 27.0]
  Responders: post-cetuximab MP-1 alpha | 7.0 [4.0 to 11.0]
  Non-responders: post-cetuximab MP-1 alpha | 3.0 [2.0 to 21.0]

3. Primary Outcome: T Cell Activation
Description: T cell activation measured at pre-/post-cetuximab exposure
Time Frame: as for outcome 1
Population: Participants that received preoperative treatment with single-agent cetuximab for a minimum of 3-4 weeks.
Measure: Median (Inter-Quartile Range); unit: percentage of T cell activation
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 33
percentage of T cell activation
  Pre-cetuximab | 0.25 [0.20 to 0.30]
  Post-cetuximab | 1.0 [0.90 to 1.40]

4. Secondary Outcome: Frequency of EGFR-specific T Cells (EGFR853-861 Peptide-specific Tetramer+ CD8+T Cells)
Description: Difference in frequency of circulating EGFR-specific T cells between cetuximab-treated and cetuximab-naive patients
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: EGFR+ T cells/10^4 T cells
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 39
EGFR+ T cells/10^4 T cells
  no cetuximab-treatment | 45 [0 to 150]
  cetuximab-treatment | 120 [0 to 300]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time during and after study treatment that participants lived with disease that did not progress per RECIST 1.0. Progression per RECIST 1.0 is defined as a 20% increase the in longest dimension (LD) lesion from Nadir.
Time Frame: Up to 54 months
Measure: Median (Full Range); unit: months
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 40
months | 24 [1 to 54]

6. Secondary Outcome: Overall Survival (OS)
Description: Number of patients remaining alive.
Time Frame: Up to 2 years
Population: All patients enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 40
participants | 40

7. Secondary Outcome: Objective Response (Rate)
Description: The percentage of participants that experienced a response to study treatment, per RECIST 1.0: Number of participant with (Complete Response (CR) + number of participants with Partial Response (PR) / Total number of participants evaluable for response.
Time Frame: Up to 2 years
Population: Participant that where evaluable for response to treatment with cetuximab (400 mg/m2 then 250mg/m2/week) for 3-4 weeks preoperatively, followed by adjuvant chemoradiation with or without cetuximab.
Measure: Number; unit: percentage of participants
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 33
percentage of participants | 33

8. Secondary Outcome: 3-year Progression-free Survival (PFS)
Description: Percentage of participants alive at 3 years that did not experience disease progression per RECIST 1.0. Progression per RECIST 1.0 is defined as a 20% increase the in longest dimension (LD) lesion from Nadir.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 40
percentage of participants | 84 [71 to 98]

9. Secondary Outcome: Change in Tumor Size
Description: Largest percent change (decrease) in tumor size before and after neoadjuvant cetuximab.
Time Frame: as for outcome 1
Measure: Number; unit: percent
Arm/Group | Neo-Adjuvant Cetuximab
Number analyzed (Participants) | 16
percent | 10

ADVERSE EVENTS:
Arm/Group | Neo-Adjuvant Cetuximab
All-Cause Mortality (participants affected / at risk) | 32/40
Serious Adverse Events (participants affected / at risk) | 8/40
Other Adverse Events (participants affected / at risk) | 32/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neo-Adjuvant Cetuximab (N=40)
Hypothyroidism (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Mania (Psychiatric disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neo-Adjuvant Cetuximab (N=40)
Anemia (Blood and lymphatic system disorders) | 15
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Dry eye (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 18
Esophageal pain (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 11
Mucositis oral (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 13
Oral pain (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 3
Edema face (General disorders) | 2
Fatigue (General disorders) | 13
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 2
Pain (General disorders) | 9
Infections and infestations - Other, specify (Infections and infestations) | 6
Skin infection (Infections and infestations) | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 6
Cholesterol high (Investigations) | 4
Creatinine increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 3
Lymphocyte count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 5
Weight loss (Investigations) | 19
White blood cell decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 9
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 16
Anxiety (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 6
Renal calculi (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 19
Hypertension (Vascular disorders) | 10
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes